CLINICAL TRIAL: NCT02279732
Title: A Randomized, Multicenter, Double-Blind, Multinational, Phase 3 Trial Comparing the Efficacy of Ipilimumab in Addition to Paclitaxel and Carboplatin Versus Placebo in Addition to Paclitaxel and Carboplatin in Subjects With Stage IV/Recurrent Non-Small Cell Lung Cancer (NSCLC) With Squamous Histology
Brief Title: Phase 3 Trial in Squamous Non Small Cell Lung Cancer Subjects Comparing Ipilimumab Plus Paclitaxel and Carboplatin Versus Placebo Plus Paclitaxel and Carboplatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA184-153; 2014-002604-25 (EudraCT Number)
Record Dates: First submitted 2014-10-14; First posted 2014-10-31 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-07

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Paclitaxel; BMS 181339; Carboplatin; Ipilimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: Carboplatin + Paclitaxel + Ipilimumab (Experimental): Paclitaxel 175 mg/m² IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by modified WHO (mWHO)
  Carboplatin Area Under the Curve (AUC6) IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by mWHO
  Ipilimumab 10 mg/kg IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by mWHO
  Interventions: Biological: Paclitaxel; Biological: Carboplatin; Biological: Ipilimumab
- Arm 2: Carboplatin + Paclitaxel + Placebo (Experimental): Carboplatin AUC6 IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by mWHO
  Paclitaxel 175 mg/m² IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by mWHO
  Placebo IV Solution Every 3 weeks during induction and every 12 weeks during maintenance until disease progression declared by mWHO
  Interventions: Biological: Paclitaxel; Biological: Carboplatin; Other: Placebo

INTERVENTIONS:
Biological: Paclitaxel
  Other Names: Taxol®; BMS-181339
Biological: Carboplatin
  Other Names: Paraplatin®
Biological: Ipilimumab
  Other Names: MDX-010; BMS-734016
  Arms: Arm 1: Carboplatin + Paclitaxel + Ipilimumab
Other: Placebo — 0.9% sodium chloride injection, USP, or 5% dextrose injection
  Arms: Arm 2: Carboplatin + Paclitaxel + Placebo

SUMMARY:
The purpose of the study is to determine whether Ipilimumab plus Paclitaxel and Carboplatin will extend the life of patients with squamous only non small cell lung cancer more than placebo plus Paclitaxel and Carboplatin.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Subjects with NSCLC of predominantly squamous histology documented by histology or cytology from brushing, washing or needle aspiration of a defined lesion but not from sputum cytology alone
* Stage IV or Recurrent NSCLC (per the 7th International Association for the Study of Lung Cancer (IASLC) classification)
* At least 1 measurable tumor lesion, as defined by mWHO criteria, that is not located in a previously irradiated area
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1

Exclusion Criteria:

* Brain metastases
* Malignant pleural effusion that is recurrent
* Documented history of severe autoimmune or immune mediated symptomatic disease that required prolonged (more than 2 months) systemic immunosuppressive (ie, steroids) treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (35):
- China (18):
  - Local Institution, Beijing, Beijing Municipality
  - Local Institution, Chongqing, Chongqing Municipality
  - Local Institution, Fuzhou, Fujian
  - Local Institution, Guangzhou, Guangdong
  - Local Institution, Shantou, Guangdong
  - Local Institution, Zhengzhou, Henan
  - Local Institution, Changsha, Hunan
  - Local Institution, Nanjing, Jiangsu
  - Local Institution, Changchun, Jilin
  - Local Institution, Xi'an, Shan3xi
  - Local Institution, Shanghai, Shanghai Municipality
  - Local Institution, Chengdu, Sichuan
  - Local Institution, Hangzhou, Zhejiang
  - Local Institution, Beijing
  - Local Institution, Chongqing
  - Local Institution, Fuzhou
  - Local Institution, Kunming
  - Local Institution, Shanghai
- Germany (6):
  - Local Institution, Berlin
  - Local Institution, Halle
  - Local Institution, Hamburg
  - Local Institution, Leipzig
  - Local Institution, Löwenstein
  - Local Institution, Mainz
- Hungary (3):
  - Pulmonologiai Klinika, Budapest
  - Csongrad Megyei Onkormanyzat Mellkasi Betegsegek Szakkorhaza, Deszk
  - Torokbalinti Tudogyogyintezet, Törökbálint
- Poland (3):
  - Oddzial Onkologiczny, Elblag
  - Oddzial Chemioterapii, Poznan
  - Klinika Nowotworow Pluca i Klatki Piersiowej, Warsaw
- Local Institution, Singapore, Singapore
- South Korea (4):
  - Local Institution, Cheongju-si, Chungcheonbuk-do
  - Local Institution, Suwon, Gyeonggi-do
  - Local Institution, Hwasun-gun, Jeollanam-do
  - Local Institution, Seoul

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 342 participants enrolled, 295 were randomized to ipilimumab (148) and placebo arms (147). After chemotherapy, double blinded study treatment, which was the focus of the study, was started.Of all randomized participants, only 98 (ipilimumab arm) and 106 (placebo arm) participants received at least one dose of blinded study therapy.
Groups:
- Ipi + PAC/CAR: Ipilumumab + paclitaxel/Carboplatin
- Placebo + PAC/CAR: Placebo + Carboplatin/Paclitaxel
Period: Overall Study
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR
Started (Started = Participants treated with double blind therapy) | 98 | 106
Completed (Completed) | 0 | 0
Not Completed | 98 | 106
Not completed — Death | 23 | 20
Not completed — Disease Progression | 13 | 3
Not completed — Withdrawal by Subject | 2 | 7
Not completed — Adverse Event | 1 | 2
Not completed — Administrative Reason By Sponsor | 0 | 2
Not completed — Study Drug Toxicity | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Maximum Clinical Benefit | 1 | 0
Not completed — Subject Requested to Discontinue | 0 | 1
Not completed — Other | 53 | 67
Not completed — Other | 3 | 3

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of blinded study therapy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR | Total
Number analyzed (Participants) | 98 | 106 | 204
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.9 (6.89) | 59.8 (8.22) | 60.3 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
  Male | 87 | 93 | 180
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 81 | 80 | 161
  Non-Chinese | 17 | 26 | 43

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) of All Randomized Participants Who Received at Least One Dose of Blinded Study Therapy
Description: OS is defined as the time from the date of randomization until the date of death. For those participants who have not died, OS was censored on the last date the participant was known to be alive.
Time Frame: Approximately 43 months post study start
Population: All participants who were randomized and received at least 1 dose of blinded study therapy.The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, no data was collected for this primary endpoint
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR
Number analyzed (Participants) | 98 | 106
months | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, the primary endpoint was not analyzed for study CA184-153 | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, the primary endpoint was not analyzed for study CA184-153

2. Secondary Outcome: Overall Survival of All Randomized Participants
Description: as for outcome 1
Time Frame: Approximately 43 months post study start
Population: All participants who were randomized to a treatment arm. The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, no data was collected for this secondary endpoint
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR
Number analyzed (Participants) | 148 | 147
months | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184153 effective 25-Sep-2015. As a result, the primary endpoint was not analyzed for study CA184-153 | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184153 effective 25-Sep-2015. As a result, the primary endpoint was not analyzed for study CA184-153

3. Secondary Outcome: Progression-free Survival (PFS) Among All Randomized Particiapants Who Received at Least One Dose of Blinded Study Therapy Using Modified World Health Organization (mWHO) Criteria
Description: PFS is defined as the time between the date of randomization and the date of progression per mWHO criteria or death, whichever occurs first. A participant who died without reported progression per mWHO criteria was considered to have progressed on the date of death. For those participants who remained alive and had not progressed, PFS was censored on the date of last evaluable tumor assessment. For those participants who remained alive and had no recorded post-baseline tumor assessment, PFS was censored on the day of randomization.
Time Frame: Approximately 43 months post study start
Population: All participants who were randomized and received at least 1 dose of blinded study therapy.The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, no data was collected for this secondary endpoint
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR
Number analyzed (Participants) | 98 | 106
months | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, the secondary endpoint was not analyzed for study CA184-53 | NA [NA to NA] — The sponsor decided to discontinue enrollment and randomization in the study CA184-153 effective 25-Sep-2015. As a result, the secondary endpoint was not analyzed for study CA184-153

ADVERSE EVENTS:
Time Frame: From first dose of blinded study therapy to 90 days after last dose of blinded study therapy (Approximately 43 months assessed up to May 2018)
Arm/Group | Ipi + PAC/CAR | Placebo + PAC/CAR
All-Cause Mortality (participants affected / at risk) | 15/98 | 9/106
Serious Adverse Events (participants affected / at risk) | 40/98 | 33/106
Other Adverse Events (participants affected / at risk) | 91/98 | 87/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipi + PAC/CAR (N=98) | Placebo + PAC/CAR (N=106)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Nodal arrhythmia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 1 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 1 | 0
Secondary hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Death (General disorders) | 1 | 1
General physical health deterioration (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 2
Sudden cardiac death (General disorders) | 1 | 0
Bacterial toxaemia (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 4 | 0
Pneumonia (Infections and infestations) | 6 | 2
Glomerular filtration rate decreased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Influenza a virus test positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4
Cerebellar ischaemia (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ipi + PAC/CAR (N=98) | Placebo + PAC/CAR (N=106)
Anaemia (Blood and lymphatic system disorders) | 34 | 35
Erythropenia (Blood and lymphatic system disorders) | 11 | 8
Leukopenia (Blood and lymphatic system disorders) | 35 | 42
Lymphopenia (Blood and lymphatic system disorders) | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 36 | 47
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 30
Constipation (Gastrointestinal disorders) | 11 | 10
Diarrhoea (Gastrointestinal disorders) | 21 | 11
Nausea (Gastrointestinal disorders) | 11 | 17
Vomiting (Gastrointestinal disorders) | 10 | 9
Asthenia (General disorders) | 6 | 9
Chest pain (General disorders) | 4 | 6
Fatigue (General disorders) | 17 | 15
Pain (General disorders) | 6 | 3
Pyrexia (General disorders) | 13 | 6
Alanine aminotransferase increased (Investigations) | 14 | 15
Aspartate aminotransferase increased (Investigations) | 12 | 10
Blood albumin decreased (Investigations) | 6 | 2
Blood alkaline phosphatase increased (Investigations) | 5 | 0
Gamma-glutamyltransferase increased (Investigations) | 6 | 1
Haemoglobin decreased (Investigations) | 35 | 28
Neutrophil count decreased (Investigations) | 7 | 7
Platelet count decreased (Investigations) | 16 | 8
Red blood cell count decreased (Investigations) | 11 | 2
Weight decreased (Investigations) | 12 | 3
White blood cell count decreased (Investigations) | 14 | 15
Decreased appetite (Metabolism and nutrition disorders) | 26 | 17
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 9
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 7
Dizziness (Nervous system disorders) | 5 | 5
Hypoaesthesia (Nervous system disorders) | 12 | 7
Neuropathy peripheral (Nervous system disorders) | 7 | 3
Insomnia (Psychiatric disorders) | 7 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 0
Rash (Skin and subcutaneous tissue disorders) | 17 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT02279732/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/32/NCT02279732/SAP_001.pdf